Does an imagined movement regime improve dexterity following conservatively managed distal radius fractures in older adults? A pilot randomised controlled trial.

Date: 21st July 2017

#### **Research Proposal- Thomas Hughes**

**Title:** Does an imagined movement regime improve dexterity following conservatively managed distal radius fractures in older adults? A pilot randomised controlled trial.

#### Introduction:

Distal radius fractures, (DRFs) are common, estimated at 71,000 a year in Britain in a prospective, multi-centred survey undertaken in 1997/8, (O'Neill et al., 2001). A recent literature review, (MacIntyre and Dewan, 2016), suggests that DRF frequency appears to be increasing worldwide.

A survey undertaken in Nottingham, (Moore and Leonardi-Bee, 2008), reported that at 1 year following DRF 63% of subjects had pain, 11% had moderate to very severe pain, (visual analogue scale). The same study reported 95% of subjects had some functional difficulty, 16% moderate to very severe difficulty, as measured with the disabilities of the arm shoulder and hand (DASH), outcome measure. This suggests that some patients may encounter some problems in recovery following this injury.

The incidence of complex regional pain syndrome, (CRPS) in the conservatively managed DRF population has been reported as 32.2%, (Jellad, Salah and Frih, 2014). This study uses recognised criteria for diagnosing CRPS which gives the reader increased confidence that the diagnosis is correct, (Laver-Fawcett, 2007).

In a rigorous, systematic Cochrane review, (O'Connell et al., 2013), a graded motor imagery programme is suggested to reduce pain and improve function in adults with CRPS. It is further suggested that the somatosensory cortex, (SSC) is negatively affected by CRPS, (Di Pietro et al. 2013), and that imagery programmes, (which include imagined movements), may positively influence the SSC, (Moseley, 2004 and Priganc and Stralka, 2011).

It has been reported in several non-randomised controlled trials that immobilisation of the upper limb in healthy individuals may negatively affect the SSC. This was illustrated by reduced tactile perception and reduced activation of the SSC, (Lissek et al., 2009), and impaired laterality recognition, (Toussaint and Meugnot, 2013, Meugnot et al., 2015 and Meugnot and Touissaint, 2015). Decreased cortical excitability has been demonstrated using trans-cranial magnetic stimulation and electromyography in non-randomised controlled trial, (Kaneko et al., 2003), where eight orthopaedic patients, (injuries not recorded), were immobilised in a DRF-type cast and compared to healthy individuals. Changes in intra-cortical inhibition and facilitation were demonstrated in a small study investigating 9 immobilised subjects with distal radius fractures, (Zanette et al., 2004). These changes could demonstrate a change in the SCC. A small, pilot randomised controlled trial, (RCT), (Frenkel et al., 2014), immobilised healthy individuals for three weeks and found that 15 minutes of imagined wrist movement each day preserved wrist extension and ulnar deviation range of motion. The authors recommend that imagined movement should be studied in orthopaedic rehabilitation.

No studies investigating imagined movements in subjects with distal radius fracture were identified in a search using a systematic approach, (appendix 1). There are two current studies, (Broekstra and Stenekes, 2015 and Schott and Korbus, 2014), that are investigating imagined movements in the distal radius population but these have yet to be published. The methodology and the exact motor imagery programmes for the intervention group are unclear. One commonality is that both studies are only using female subjects. When examining the local metrics at Aneurin Bevan University Health-Board, (ABUHB), approximately 20% of this population are male. It is suggested that although relatively small, this group should be included to more closely represent the population of interest. It is suggested that this could be addressed in this proposed study.

The Purdue pegboard was designed to assess manipulative dexterity, (Tiffin and Asher, 1948). In a systematic review the Parkinson evidence database to guide

effectiveness task force, (Kegelmeyer et al., 2014), recommends the Purdue pegboard to measure fine motor activity and dexterity in Parkinson's disease. Its application in assessing the dexterity of neurologically impaired subjects suggests it is suitable for use in this trial as a measure of motor control/ SSC function.

In summary, it is suggested that DRFs are common and immobilisation for conservative treatment may cause changes in the SSC. The SSC may be positively influenced by imagined movements. No studies were identified which investigate this topic using recognised outcome measures for pain and dexterity.

#### **Study Objectives**

The aim is to undertake a pilot RCT to investigate whether an imagined movement regimen improves dexterity in conservatively managed DRFs in adults over 50, when compared to control.

#### Other objectives are:

- 1) To assess dexterity using the Purdue pegboard in adults over 50 years old with conservatively managed DRFs, following an imagined movement regimen when compared to control.
- 2) To evaluate pain using a visual analogue scale, (VAS) in adults over 50 years old with conservatively managed DRFs, following an imagined movement regimen when compared to control.
- 3) To evaluate active range of motion using goniometry in adults over 50 years old with conservatively managed DRFs, following an imagined movement regimen when compared to control.
- 4) To test research procedures in the same study, and highlight any specific problems.

#### **Study Plan**

#### <u>Design</u>

When examining a new treatment, a randomised controlled trial can be considered to produce the best level of evidence, (Aveyard, 2014). Randomising reduces selection bias and increases the chances of the control and intervention groups being similar to each other, (May, 2011 and Denscombe, 2010). Controlling the extraneous variables, and having a control group attempts to isolate the intervention and its relationship on outcome, (Bowling, 2014). Due to costs the assessor cannot be blinded to the group allocation. This is recognised as a potential source of bias but is unavoidable in this pilot study.

#### Sample

Subjects will be recruited from two of the local Accident and Emergency departments on their initial visit with DRF. The inclusion and exclusion criteria are tabulated in appendix 2.

#### Number of participants:

It is difficult to predict how many participants will be available that meet the criteria. An aim of this pilot study is to test procedure, this includes recruitment. Generally it's preferable to have more subjects in a study, (Blaxter, Hughes and Tight, 2010), however the numbers need to be manageable, (Denscombe 2010). Metrics from the two sites between April and September 2016 shows an average of 33 patients with DRF over the age of 50 per month. There tends to be a higher frequency of DRF due to falls in the winter months, (MacIntyre and Dewan, 2016), therefore this may be a conservative estimate. If we allow for subjects declining to participate or not meeting criteria, (estimate 25%), and factor in a drop-out rate of 20%, (drop-out rates reported to be over 20% in 18% of RCTs, Wood, White and Thompson, 2004), this could result in a sample size of approximately 20 per month. If recruitment runs for 2 months, (see appendix 3), that could lead to approximately 40 subjects, 20 in each group.

#### **Procedures:**

See appendix 4 for flow chart of how subjects move through the study.

At initial attendance in Accident and Emergency, subjects that meet the inclusion criteria will be offered an information sheet, (appendix 5) and will be asked whether they want to be included in the trial. If they agree, a consent form regarding being contacted about the study, (appendix 6), and an assessment form, (appendix 7) will be completed by the advanced nurse practitioner. The forms will be given to the primary researcher and filed securely to comply with The Data Protection Act, (1998). All patients, including those who do not wish to participate or don't meet the criteria will be given the standard advice and exercise booklet, (appendix 8 without italic section). This is usual for this group of patients.

The lead researcher will contact each subject within 3 days to discuss the study, and arrange an appointment at 7-10 days to begin the study. This is necessary ethically in order to provide a 'cooling-off' period for the subjects to consider whether they wish to participate. It will also give time for radiology reports to be completed and any subjects with discounted radius fracture can be excluded.

Potential subjects attending the initial appointment at 7-10 days will be offered the full consent form, (appendix 9). Those that do not attend or do not consent will be referred back to Accident and Emergency and return to usual care. Those that consent will be randomised into control or intervention group using a computerised random number generator. The control group will continue with maintenance exercises. The intervention group will have the same exercises as the control group plus imagined wrist exercises, (appendix 8 including italic section). The exercises will be taught to the subject by reading through the booklet with them, this ensures the advice is standardised. As the intervention is targeting the SSC, high frequency is considered important, (Magill and Anderson, 2014). The imagined movement programme, is amalgamated from that described by Moseley (2004) and Frenkel et al., (2014), and will consist of imagined wrist movement in all planes. The frequency of 15 minutes every waking hour, (Moseley, 2004), is deemed impractical and, as previously mentioned, 15 minutes of mental practice a day preserved range of motion, (Frenkel et al., 2014). Therefore approximately 10-15 minutes, four times a day has been selected as a pragmatic compromise and mirrors routine advice.

An appointment will be arranged as soon as is practically possible, aiming for the same day or day after removal of plaster at approximately 4-8 weeks, (varies between teams). This is to reduce the chance of movement out of plaster affecting the outcome measures.

#### **Outcome Measures**

The primary outcome measures of dexterity using the Purdue peg-board, and secondary outcome measures of pain and active wrist range of motion will be measured and recorded, (see appendix 10). The Purdue peg-board will be used as per standardised procedure, (Lafayette, 2002). It has established reliability and validity, (albeit not in this specific population, Yancosek and Howell, 2009), and normative data, (Tiffin and Asher, 1948). It is used in this study to measure fine finger-tip dexterity which could be influenced by changes in the SSC. The Visual Analogue Scale for pain is widely used in research and clinical trials to measure pain, (Paul-Dauphin, 1999) and has reported reliability in a range of patient groups including acute pain, (Bijur, Silver and Gallagher, 2001). Goniometry is widely used in research to measure joint movements and has reported reliability and validity, (Gajdosik and Bohannon, 1987, Horger, 1990, and Carter et al., 2009).

.

#### <u>Analysis</u>

Demographic data will be correlated and compared across groups using descriptive statistics, (Blaxter, Hughes and Tight, 2010). The data will be compared using inferential statistics to establish whether the groups were similar, (Denscombe, 2010). The outcome measures being used produce ordinal/ratio data and inferential statistics will be used to see if there is a difference between the control and intervention groups. It is recognised that the sample size will be too small to determine statistical significance, (Suresh and Chandrashekara, 2012), but the study will collect data and test processes that could be used in a full study.

#### **Ethics**

Benefits and risks are included in the participant information sheet, (appendix 5). The subjects will be fully informed of the intervention, their commitment and that they can leave at any time. Subjects who do not consent will be discharged from the study and return to usual care through accident and emergency. Usual care is that patients are normally referred to physiotherapy after removal of plaster, (it is worth noting that some patients are not referred). All subjects will have 2 additional appointments compared to usual care, one at day 7-10, and one for their final assessment. This will incur time and costs to each subject, but it may benefit them as they will see a Physiotherapist and could discuss any concerns and have their exercises reinforced. Subjects will also commence their physiotherapy treatment approximately 1 week earlier than usual which may be seen as a benefit. The subject is informed of this in the information sheet.

University of Derby Health and Social Care Research Ethics Committee have approved the proposal and this proposal is being submitted as part of the IRAS process for NHS REC approval.

#### References.

Aveyard, H. (2014) *Doing a literature review in health and social care: a practical quide.* 3<sup>rd</sup> Edition. Maidenhead: McGraw-Hill Open University Press.

Bijur, P.E., Silver, W. and Gallagher, J. (2001) 'Reliability of the Visual Analog Scale for Measurement of Acute Pain', *Academic Emergency Medicine* 8 (12): pp 1153-1157.

Blaxter, L., Hughes, C., and Tight, M. (2010). *How to Research.* 4<sup>th</sup> Edition. Maidenhead: McGraw-Hill Open University Press.

Bowling, A. (2014) *Research methods in health: investigating health and health services.* 4<sup>th</sup> Edition. Maidenhead: McGraw-Hill Open University Press.

Broekstra, D.C., and Stenekes, M.W., (2015) 'Motor Imagery in Rehabilitation After a Distal Radius Fracture (MIDRF)', *Clinical Trials.gov* Available at https://clinicaltrials.gov/ct2/show/NCT01921062 (Accessed 10<sup>th</sup> October 2016).

Carter, T.I., Pansy, B., Wolff, A.L., Hillstrom H.J., Backus, S.I., Lenhoff, M. and Wolfe, S.W. (2009) 'Accuracy and reliability of three different techniques for manual goniometry for wrist motion: a cadaveric study', *Journal of Hand Surgery (American)* 34 (8) pp1422-1428.

Denscombe, M. (2010) *The good research guide: for small-scale social research projects*. 4<sup>th</sup> Edition. Maidenhead: McGraw-Hill Open University Press.

Di Pietro, F., McAuley, J.H., Parkitny, L., Lotze, M., Wand, B.M., Moseley, L. and Stanton, T.R. (2013) 'Primary Somatosensory Cortex Function in Complex Regional Pain Syndrome: A Systematic Review and Meta-Analysis', *Journal of Pain* Vol. 14, Issue 11, pp 1270-1288.

Frenkel, M.O., Herzig, D.S., Gebhard, F., Mayer, J., Becker, C., and Einsiedel, T. (2014) 'Mental practice maintains range of motion despite forearm immobilization: A pilot study in healthy persons', *Journal of Rehabilitative Medicine* 46: pp 225-232.

Gajdosik R.L. and Bohannon, R.W. (1987) 'Clinical measurement of range of motion: Review of goniometry emphasizing reliability and validity', *Physical Therapy* 67 (12) pp 1867-1872.

Horger M.M. (1990) 'The reliability of goniometric measurements of active and passive wrist motions', *American Journal of Occupational Therapy* 44(4): pp 342-348.

Jellad, A., Salah, S. and Frih, Z.B.S. (2014) 'Complex Regional Pain Syndrome Type I: Incidence and Risk Factors in Patients With Fracture of the Distal Radius', *Archives of Physical Medicine and Rehabilitation* 95 pp 487-92.

Kaneko, F., Murakami, T., Onari, K., Kurumadani, H., and Kawaguchi, K. (2003) 'Decreased cortical excitability during motor imagery after disuse of an upper limb in humans', *Clinical Neurophysiology* 114 pp 2397-2403.

Kegelmeyer, D., Ellis, T., Esposito, A., Gallagher, R., Harro, C., Hoder, J., Hussey, E., Oneal, S., (2014) 'Parkinson EDGE task force recommendations by disease stage' http://www.neuropt.org/docs/default-source/parkinson-edge/pdedge-all-documents-combined.pdf?sfvrsn=2 Accessed 9<sup>th</sup> December 2016.

Lafayette, (2002) *Purdue Pegboard Test: User Instructions* USA: Lafayette Instrument Group.

Laver-Fawcett, A. (2007). "Standardisation and Test Development." In: Laver-Fawcett, A. (ed) *Principles of assessment and outcome measurement for Occupational Therapists and Physiotherapists: theory, skills and application.* Chichester: John Wiley and Sons; pp 151-168.

Lissek, S., Wilimzig, C., Stude, P., Pieger, B., Kalisch, T., Maier, C., Peters, S.A., Nicolas, V., Tegenthoff, M. and Dinse, H.R. (2009) 'Immobilization Impairs Tactile Perception and Shrinks Somatosensory Cortical Maps', *Current Biology* 19 pp 837-842.

MacIntyre, N.J. and Dewan, N. (2016) 'Epidemiology of distal radius fractures and factors predicting risk and prognosis', *Journal of Hand Therapy*, 29: pp 136-145.

Magill, R.A. and Anderson, D. (2014) *Motor Learning and Control: Concepts and Applications*. 10<sup>th</sup> Edition. New York: McGraw-Hill Education

May, T. (2011) *Social research: issues, methods and process.* 4<sup>th</sup> Edition. Maidenhead: Open University Press.

Mental Capacity Act 2005. Available at:

http://www.legislation.gov.uk/ukpga/2005/9/pdfs/ukpga\_20050009\_en.pdf (Accessed 1st February 2017).

Meugnot, A., Agbangla, N.F., Almecija, Y. and Toussaint, L. (2015) 'Motor imagery practice may compensate for the slowdown of sensorimotor processes induced by short-term upper-limb immobilization', *Psychological Research* 79: pp 489-499.

Meugnot, A., and Toussaint, L. (2015) 'Functional plasticity of sensorimotor representations following short-term immobilization of the dominant versus non-dominant hands', *Acta Psychologica* pp 51-56.

Moore, C.M., and Leonardi-Bee, J. (2008) 'The prevalence of pain and disability one year post fracture of the distal radius in a UK population: A cross sectional survey', *BMC Musculoskeletal Disorders* 9: 129

Moseley, G.L. (2004) 'Graded motor imagery is effective for long-standing complex regional pain syndrome: a randomised controlled trial', *Pain*. Pp 108:192–198.

O' Connell, N.E., Wand, B.M., McAuley, J., Marston, L., and Moseley, G.L. (2013) 'Interventions for treating pain and disability in adults with complex regional pain syndrome- an overview of systematic reviews (Review)', *Cochrane Database of Systematic Reviews* Issue 4.

O'Neill, T.W., Cooper, C., Finn, J.D., Lunt, M., Purdie, D., Reid, D.M., Rowe, R., Woolf, A.D. and Wallace, W.A. (2001) 'Incidence of Distal Forearm Fracture in British Men and Women', *Osteoporosis International* 12: pp 555-558.

Paul-Dauphin, A., Guillemin, F., Virion, J.M and Briancon, S. (1999) 'Bias and Precision in Visual Analogue Scales: A Randomized Controlled Trial', *American Journal of Epidemiology* 150 (10) pp 1117-1127.

Priganc, V.W., and Stralka, S.W. (2011) 'Graded motor imagery', *Journal of Hand Therapy* 24: pp 164–168.

Schott, N., and Korbus, H. (2014) 'Preventing functional loss during immobilization after osteoporotic wrist fractures in elderly patients: a randomized clinical trial', *BMC Musculoskeletal Disorders* 15: 287.

Suresh, K.P., and Chandrashekara S. (2012) 'Sample size estimation and power analysis for clinical research studies', *Journal of Human Reproductive Sciences* 5 (1): pp 7-13.

The Data Protection Act 1998. Available at:

http://www.legislation.gov.uk/ukpga/1998/29/contents (Accessed 10<sup>th</sup> October 2016).

Tiffin, J. and Asher, E.J. (1948) 'The Purdue Pegboard: norms and studies of reliability and validity', *Journal of Applied Psychology* 32: pp 234-247.

Toussaint, L., and Meugnot, A. (2013) 'Short-Term Limb Immobilization Affects Cognitive Motor Processes', *Journal of Experimental Psychology: Learning, Memory and Cognition* 39 (2) pp 623-632.

Wood, A.M., White, I.R., and Thompson, S.G. (2004) 'Are missing outcome data adequately handled? A review of published randomized controlled trials in major medical journals', *Clinical Trials* 1: pp 368-376.

Yancosek, K.E. and Howell, D. (2009) 'A narrative review of dexterity assessments', *Journal of Hand Therapy* 22: pp 258-270.

Zanette, G., Manganotti, P., Fiaschi, A. and Tamburin, S. (2004) 'Modulation of motor cortex excitability after upper limb immobilization', *Clinical Neurophysiology* 115: pp 1264-1275.

#### Appendix 1. Literature search strategy.

Subject terms: ("motor imagery" OR imagined OR mental OR thought OR think) AND (hand OR wrist) AND (all text) (immobilisation OR static OR plaster OR splint OR fracture) NOT (CRPS OR "complex regional pain").

When fracture OR radius was added, no further articles were identified, it was therefore omitted from the search and the research question for this review became, does motor imagery/imagined movement improve outcome following wrist immobilisation?

#### Inclusion criteria:

- Any article that explores the use of motor imagery/imagined movements with immobilised hand/s or wrist/s
- Written in English language.
- Human.
- Published in a peer reviewed journal.

#### Exclusion criteria:

- Not English language.
- Any article not exploring the use of motor imagery/imagined movements with immobilised hand/s or wrist/s.
- Not human.

#### Date published

No date restrictions are applied as all articles identified are published since 1990 and as only 49 articles were identified in total it was not deemed necessary to limit by date and risk missing key articles.

#### <u>Databases</u>

Library plus and Google scholar

#### **Further Searching**

In addition to the database and journal searches, the reference lists of the identified articles and any previous work by the authors were scrutinised using the same inclusion and exclusion criteria.



Abstracts scrutinised and articles not meeting inclusion criteria, (n=73), removed.

#### 6 articles

Bassolino et al., (2013), Frenkel et al., (2014), Meugnot et al., (2015), Meugnot et al., (2016), Schott and Korbus, (2014), Stenekes et al., (2009).



References scrutinised and authors' previous work searched, 2 further articles identified, including 1 unpublished, current trial, the authors were contacted, no information available yet.

8 articles (those above plus)
Schott et al., (2013), Broekstra and Stenekes, (current trial)

## Appendix 2. Inclusion and exclusion criteria and justification.

| Inclusion Criteria | Justification/Reason |
|---|---|
| Age > 50 | Used commonly in research, (MacIntyre and |
| | Dewan, 2016). |
| | Avoids the variable of relatively high velocity |
| | injuries sustained by the younger population |
| | influencing outcome. |
| Closed distal radius fracture | Population of interest. |
| | Prevents possible impact of other variables |
| | for example wound, infection, operative |
| | input. |
| Lives within ABUHB geographically | If subject lives outside of ABUHB |
| | geographically they may not be funded for |
| | their care and would normally be referred |
| | locally for their treatment. |

| Exclusion Criteria | Justification/Reason |
|---|---|
| Age < 50 | See inclusion criteria (Age>50). |
| Lives outside ABUHB/unable to attend | Would not be able to attend for |
| appointments | intervention/assessment. |
| Open distal radius fracture | See inclusion criteria (closed distal radius |
| | fracture). |
| Subjects that require surgery | To prevent a possible impact from this |
| | variable |
| Subjects where a fracture is subsequently | Subject would no longer be in the population |
| ruled out | of interest. |
| Any additional upper limb injury | To prevent a possible impact from this |
| | variable and may prevent ability to |
| | participate in the intervention or control |
| | group. |
| Bilateral wrist fracture | Would prevent ability to participate in the |
| | intervention group as contralateral wrist is |
| | used. |
| Unable to consent | Consent required to participate. |
| (Subject lacks capacity to consent for | |
| example due to a mental health condition, | |
| learning disability, dementia or another | |
| similar condition using the Mental Capacity | |
| Act, 2005 as a guide) | |
| Unable to follow instructions or speak | Would prevent ability to participate. |
| English | |
| Pre-existing wrist injury, deformity or | To prevent a possible impact from this |
| neurological impairment of either upper | variable. Subject may not be able to |
| limb | participate. |
| Subject describes significant emotional | To reduce the subject experiencing undue |
| and/or psychological trauma at time of | stress and reduce the incidence of additional |
| injury | debriefing with these subjects which would |

| <br> |
|---------------------------------------------|
| add time to the assessments and potentially |
| add a confounding variable to the study |

#### Appendix 3. Planned time line for study, (adjusted due to extension granted)

| | July | August | Sep | Oct | Nov | Dec | Jan | Feb | March |
|---|---|---|---|---|---|---|---|---|---|
| Continue literature search and review | | | | | | | | | |
| Pilot (dependent on ethics) | | | | | | | | | |
| Recruitment | | | | | | | | | |
| Main data collection | | | | | | | | | |
| Write method section | | | | | | | | | |
| Data collation and analysis | | | | | | | | | |
| Write results section | | | | | | | | | |
| Write discussion and conclusion | | | | | | | | | |
| Complete typing, editing, binding | | | | | | | | | |

May require deferring/expediting dependent on ethical approval but time scales would remain similar.

#### Appendix 4. Flow diagram of progress through study.

#### Day 0

Potential subject attends Accident and Emergency with a distal radius fracture.

All patients are provided with an advice and exercise sheet, (appendix 8 without italic section). Advanced Practice Nurse ensures suitability with inclusion and exclusion criteria and an information sheet, (appendix 5), and a consent to be contacted form (appendix 6) are completed.

If consent is given then If consent **Patient** demographic data is not given collected using form, discharged from study and (appendix 7). returned to usual care Day 2-3 Potential subject telephoned by primary researcher. Any questions or concerns are able to be discussed. An appointment is arranged for the subject to commence the study. Consent not given Day 7-10 Subject attends initial appointment and is offered full consent form, (appendix 9). Consent given Subject randomised into control or treatment group.

Control group continue with same exercises, treatment group given additional imagined movement exercises (appendix 8 with italics) issued.

Assessment appointment arranged to correlate with removal of plaster cast.



Day 28-56 (dependent on length of immobilisation)

Assessment of primary and secondary outcome measures, (appendix 10).

Study terminates, standard physiotherapy begins.

#### Participant information sheet



#### PARTICIPANT INFORMATION SHEET

#### STUDY TITLE

Does an imagined movement regime improve dexterity following conservatively managed distal radius fractures in older adults? A pilot randomised controlled trial.

You are being invited to take part in a research study. Please take time to read the following information carefully as it is important that you understand why the research is being done and what is involved. Feel free to discuss this with your friends and family and take your time to decide. You can then decide whether or not you wish to take part.

#### WHO IS ORGANISING AND FUNDING THE RESEARCH?

I am conducting this research as part of my MSc in Hand Therapy as a student of Derby University, College of Health and Social Care. Aneurin Bevan University Health Board is supporting me in terms of my time. There is no direct funding.

#### WHAT IS THE PURPOSE OF THE STUDY?

Patients with a broken/fractured wrist can have problems with stiffness, pain and use of their hand and arm for several months following removal of plaster. This study is investigating whether imagined movements whilst in the plaster improves your dexterity and/or reduces pain and/or improves movement. It is a randomised control trial; this means that you will be placed in either a control or experimental group.

You have been asked to participate because you have a distal radius fracture, (wrist fracture) that has been treated in plaster and you are over 50 years of age.

#### DO I HAVE TO TAKE PART?

Taking part in this study is entirely optional. If you do decide to take part you will be given this information sheet to keep and be asked to sign a consent form to be contacted by phone to arrange an appointment. If you decide to take part you are free to withdraw at any time and without giving a reason. Any information collected up to the point of withdrawal will be retained. This study will not prevent you from attending any hospital or physiotherapy appointments.

#### WHAT WILL HAPPEN TO ME IF I TAKE PART?

All participants will be contacted by telephone within 3 days of joining the study to ask if you want to be involved in the study. If you do not want to be involved you will be referred back to Accident and Emergency and return to usual care which will normally involve a physiotherapy referral after removal of your plaster. If you want to be involved an appointment will be arranged for you about 1 week after you first attended Accident and Emergency. This is an extra appointment that you would not normally have. At this appointment you will see the lead researcher who is a Clinical Specialist Physiotherapist and be asked to fill in a consent form. If you do not want to be involved you will be referred back to Accident and Emergency and return to usual care, (as described earlier). If you agree to take part you will be put into one of two groups. One group, the control group, will be taught the usual exercises to maintain the shoulder, elbow and finger movements whilst in plaster. The other group, the experimental group, will have the same exercises and some additional exercises where you imagine moving your wrist whilst it is still in plaster. Both groups will be asked to do these exercises 4 times a day. It is anticipated they will take you no more than 15 minutes each time.

A final assessment appointment will be arranged soon after your plaster is removed. At this appointment the lead researcher will measure your wrist movements, (as an angle), your pain level, (using a line scale), and your ability to manipulate small objects using a pegboard, which involves placing small pegs into holes. This should take no more than 30 minutes. These appointments can only be arranged at the Royal Gwent Hospital, Newport. This will be the end of the trial for you but you will continue to attend physiotherapy as necessary.

#### WHAT ARE THE POSSIBLE DISADVANTAGES AND RISKS OF TAKING PART?

As mentioned previously, you will need to attend two appointments, each lasting no more than 30 minutes. These appointments are extra compared to usual care. Unfortunately there is no funding available for your travel or time. There is no cost to park at the hospital but parking is limited.

You may be randomised to the control group; this means that you will receive the usual exercises rather than the treatment being investigated.

There are no known risks associated with the two exercise plans.

Measuring your wrist movements and dexterity may be uncomfortable but will not be harmful as we would normally encourage early movement when the plaster is removed.

#### WHAT ARE THE POSSIBLE BENEFITS OF TAKING PART?

There are no intended clinical benefits to taking part in the study however you will attend physiotherapy slightly earlier than normal, this may give you the chance to ask any questions and raise any concerns you may have.

If you are in the control group you will still receive the usual exercises to ensure you are not penalised for participating.

Research is essential in ensuring we use evidence to guide our treatment. By participating you may help to improve our understanding of this topic and possibly improve future patient care.

#### WILL MY DETAILS BE KEPT CONFIDENTIAL?

All information collected will be kept strictly confidential, (subject to legal limitations).

Your G.P. and/or consultant will be informed if you decide to participate. Your details will be anonymised and all data will be securely stored either in locked cabinets or on a password protected computer. No personal information will be included in the writing of this study.

#### WHAT SHOULD I DO IF I WANT TO TAKE PART?

If you want to take part please sign the consent form so that I can contact you by phone. I will phone you within three days of your plaster being applied and you will be asked again if you are happy to take part. At the first appointment you will be asked to complete a full consent form.

#### WHAT WILL HAPPEN TO THE RESULTS OF THE RESEARCH STUDY?

The results of this study will be used as my dissertation for an MSc in Hand Therapy at the University of Derby. The results of this study may be published in the form of a poster at scientific conferences, no confidential information will be used. The findings may be used to guide further study which could be published in a scientific journal, if you wish to view the results please contact me using the details below.

#### WHO HAS REVIEWED THE STUDY?

The research has been approved by the University of Derby and NHS ethics boards.

#### **CONTACT FOR FURTHER INFORMATION**

Researcher: Tom Hughes Clinical Specialist Physiotherapist, Royal Gwent Hospital, Cardiff Road, Newport NP20 2UB (01633 234491) Email tom.hughes@wales.nhs.uk

If you have any concerns about how this research is being undertaken please contact my supervisor, Sue Kennedy, Lecturer, University of Derby, College of Health and Social Care, Kedleston Road, Derby. DE22 1GB Email S.Kennedy@derby.ac.uk

THANK YOU FOR TAKING THE TIME TO READ THIS INFORMATION SHEET.

#### DATE

Version 2-17



#### RESEARCH ETHICS: CONSENT TO BE CONTACTED FORM

Does an imagined movement regime improve dexterity following conservatively managed distal radius fractures in older adults? A pilot randomised controlled trial.

#### Name, position and contact address of Researcher:

Mr Tom Hughes, Clinical Specialist Physiotherapist, (hands). Physiotherapy hand unit, physiotherapy department. Royal Gwent Hospital Cardiff Road Newport NP20 2UB

Email: tom.hughes@wales.nhs.uk

| | | | Please Initial Box |
|---|---|---|---|
| 1. | I confirm that I have read an sheet for the above study and ask questions. | | |
| 2. | I agree to be telephoned to disc<br>study and to arrange an appoin | | |
| Name | of Participant | Date | Signature |
| Name | of Researcher/Staff | <br>Date | Signature |

# Appendix 7. Baseline demographic data form.





| Subject Name |
|------------------------------------|
| Subject Hospital number |
| Date of A&E attendance |
| Subject Date of Birth |
| Subject Contact Telephone number/s |

This provides enough information to ensure the correct subject is identifiable whilst not collecting unnecessary data.



# Aneurin Bevan University Health Board Physiotherapy Directorate

# Physiotherapy advice and exercise booklet:

Wrist fractures.

This booklet gives you advice on helping your wrist to recover following a wrist fracture/break. Whilst in your plaster there are some exercises you can do which may reduce stiffness and pain.

### **Swelling and pain**

When you break your wrist it is normal to have swelling and pain. You should keep your hand elevated as much as possible. This should help with the swelling.

You may have been prescribed pain killers by a member of staff in accident and emergency. If you have any concerns or feel your pain is not under control, speak to your G.P. or pharmacist.

#### **Exercises**

It is very important to exercise, even when your wrist is immobilised in a plaster cast. It is suggested that all of these exercises are performed 4 times a day. There is a diary at the back of this booklet for you to record when you exercise. You may also wish to set an alarm to remind you when to exercise through the day.



1) Make a fist and then straighten your fingers. Repeat 10 times.



2) Make a hook/claw grip (the main knuckle joints straight with the smaller finger joints bent). Then straighten your fingers. Repeat 10 times.



3) Bring your arm forwards so that your hand goes above your head, then lower your hand. Repeat 10 times.



4) Leading with your thumb, bring your arm out to the side and above your head, then lower. Repeat 10 times.



5) Keep you elbows tucked into your side. Rotate your shoulders so that your hands move away from your body.

The next three exercises involve you imagining that you are moving the wrist that is in plaster. We recommend that you perform each of the exercises 3 times with your un-injured wrist so that you can see and feel how your 'normal' wrist moves. Then try to think about doing the same thing with your other wrist. You do not need to actually move your wrist in the plaster, you just need to imagine the wrist is moving. We think this may help to maintain the movement control part of your brain whilst your wrist is unable to move in the plaster cast.



Move your un-injured wrist slowly backwards and forwards 3 times. Concentrate on how the wrist moves and how it feels when it moves. Now, imagine doing the same exercise with your injured wrist 20 times.



Move your un-injured wrist slowly from side to side 3 times.
Concentrate on how the wrist moves and how it feels when it moves.
Now, imagine doing the same exercise with your injured wrist 20 times.



Keep your elbow tucked into your side. Move your un-injured wrist slowly so that the palm faces up and then down, 3 times. Concentrate on how the wrist moves and how it feels when it moves. Now, imagine doing the same exercise with your injured wrist 20 times.

(The section in italics is not included for the control group).

# **Exercise diary**

Please use this chart to help you remember to exercise. Tick the relevant box each time you complete your exercises.

| | Monday | | | | | Tuesday | | Wednesday | | | Thursday | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | morning | midday | afternoon | evening | morning | midday | afternoon | evening | morning | midday | afternoon | evening | morning | midday | afternoon | evening |
| Week 1 | | | | | | | | | | | | | | | | |
| Week 2 | | | | | | | | | | | | | | | | |
| Week 3 | | | | | | | | | | | | | | | | |
| Week 4 | | | | | | | | | | | | | | | | |
| Week 5 | | | | | | | | | | | | | | | | |
| Week 6 | | | | | | | | | | | | | | | | |

| | | Fr | iday | | Saturday | | | | Sunday | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | morning | midday | afternoon | evening | morning | midday | afternoon | evening | morning | midday | afternoon | evening |
| Week 1 | | | | | | | | | | | | |
| Week 2 | | | | | | | | | | | | |
| Week 3 | | | | | | | | | | | | |
| Week 4 | | | | | | | | | | | | |
| Week 5 | | | | | | | | | | | | |
| Week 6 | | | | | | | | | | | | |

If you have any questions about your exercises or have any concerns please contact the physiotherapy team using the details below.

Physiotherapy Hand Unit
Physiotherapy Outpatients
Royal Gwent Hospital
Cardiff Road
Newport
NP20 2UB
Tel: 01633 234491







#### **RESEARCH ETHICS: CONSENT FORM**

Does an imagined movement regime improve dexterity following conservatively managed distal radius fractures in older adults? A pilot randomised controlled trial.

#### Name, position and contact address of Researcher:

Mr Tom Hughes, Clinical Specialist Physiotherapist, (hands). Physiotherapy hand unit, physiotherapy department. Royal Gwent Hospital Cardiff Road Newport NP20 2UB

Email: tom.hughes@wales.nhs.uk

| | | | Please Initial Box |
|---|---|---|---|
| 1. | I confirm that I have read as sheet for the above study an ask questions. | | |
| 2. | I understand that my participal free to withdraw at any time, wif my data has been analysed no longer be able to withdraw. | vever, | |
| 3. | I understand my information securely | held | |
| 4. | I agree that my GP and the or my care will be informed of | I | |
| 5. | I agree to take part in the a | | |
| Name | of Participant | Signature | |
| Name | of Researcher | Signature | |

#### Appendix 10. Assessment data form.





| Subject Name | | |
|-------------------------------|------------------|---------|
| Hospital number | | |
| Subject Date of Birth | | |
| Date | | |
| Group allocation | Intervention | Control |
| Days since removal of plaster | | Days |
| Hand dominance | LEFT | RIGHT |
| Injured Hand | LEFT | RIGHT |
| Length of time in plaster | | Weeks |
| Wrist active ROM | Flexion | |
| | Extension | |
| | Radial Deviation | |
| | Ulnar Deviation | |
| | Supination | |
| | Pronation | |
| Purdue peg board score | Left | |
| | Right | |
| | Both hands | |
| | Left+Right+Both | |
| | Assembly | |
| | | 1 |

| <u>Pain score</u> | |
|---|---|
| No pain at all | Worst pain imaginable |
| (It will be checked that this line measures 10cm when printed/photocopied) | |

**Current medication**